CLINICAL TRIAL: NCT02370485
Title: Relative Bioavailability and the Effect of Food on the Bioavailability of LY2801653 in Healthy Subjects
Brief Title: A Study of LY2801653 in Healthy Participants Who Are Not Able to Have Children
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 15778; I3O-EW-JSBD (Other: Eli Lilly and Company)
Record Dates: First submitted 2015-02-23; First posted 2015-02-25 (Estimated); Last update posted 2015-06-19 (Estimated); Status verified 2015-06

CONDITIONS: Healthy
MeSH Terms: interventions — merestinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- LY2801653 Reference - Fasted (Experimental): Single oral dose of LY2801653 (Reference Formulation) administered in fasted state in one of three study periods.
  Interventions: Drug: LY2801653
- LY2801653 Test - Fasted (Experimental): Single oral dose of LY2801653 (Test Formulation) administered in fasted state in one of three study periods.
  Interventions: Drug: LY2801653
- LY2801653 Test - Fed (Experimental): Single oral dose of LY2801653 (Test Formulation) administered with a high fat meal in one of three study periods.
  Interventions: Drug: LY2801653

INTERVENTIONS:
Drug: LY2801653 — Administered orally

SUMMARY:
The purpose of this study is to evaluate how much of the LY2801653 drug is available in the body when given in 2 different formulations with and without a meal to healthy participants who are not able to have children. In addition, this study will measure how much of the drug gets into the blood stream and how long it takes the body to get rid of it. Information about any side effects that may occur will also be collected. The study will last about 27 days. Screening is required within 28 days prior to the start of the study.

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy sterile male and female participants
* Body mass index (BMI) of 18.0 to 32.0 kilograms per square meter (kg/m^2), inclusive
* Are willing and able to eat the protocol specified high-fat breakfast

Exclusion Criteria:

* Have consumed grapefruits or grapefruit-containing products, Seville oranges or Seville orange juice, star fruit, star fruit juice, or star fruit-containing products, or commercial apple or orange juice within 14 days prior to first dosing
* Regularly use known drugs of abuse and/or show positive findings on urinary drug screening
* Have donated blood of more than 500 milliliter (mL) within the last month

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2015-02; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics: Maximum Concentration (Cmax) for LY2801653 | Predose through 96 hours after administration of study drug in periods 1 and 2 and predose through 120 hours after administration of study drug in period 3
Pharmacokinetics: Area Under the Concentration Curve (AUC 0-∞) for LY2801653 | Predose through 96 hours after administration of study drug in periods 1 and 2 and predose through 120 hours after administration of study drug in period 3

SECONDARY OUTCOMES:
Pharmacokinetics: Maximum Concentration (Cmax) of LY2801653 and Major Metabolites LSN2800870 and LSN2887652 | Predose through 96 hours after administration of study drug in periods 1 and 2 and predose through 120 hours after administration of study drug in period 3
Pharmacokinetics: Area Under the Concentration Curve (AUC 0-∞) for LY2801653 and Major Metabolites LSN2800870 and LSN2887652 | Predose through 96 hours after administration of study drug in periods 1 and 2 and predose through 120 hours after administration of study drug in period 3

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Covance, Daytona Beach, Florida, United States